CLINICAL TRIAL: NCT03778242
Title: The Adjunctive Role of Temporary Uterine Packing Combined With Topical Tranexamic Acid for Reducing Blood Loss During Hemorrhagic Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Tranexamic Acid in Pregnant Women Undergoing Cesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: aswu/276/18
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; tranexamic acid; postpartum hemorrhage; oxytocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: open label Randomized Clinical Tria
Masking Description: open label Randomized Clinical Tria
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical tranexamic acid (Active Comparator): temporary uterine packing with gauze of the dimensions soaked with 2 gm tranexamic diluted in 60ml saline acid
  Interventions: Drug: Topical tranexamic acid
- normal saline (Placebo Comparator): temporary uterine packing with gauze of the dimensions soaked with 2 gm placebo to tranexamic diluted in 60ml saline acid
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Topical tranexamic acid — temporary uterine packing with gauze of the dimensions soaked with 2 gm tranexamic diluted in 60ml saline acid
  Other Names: Active Comparator
  Arms: Topical tranexamic acid
Drug: normal saline — 2 placebo ampoules to TA in 100 ml saline by slow infusion
  Other Names: Placebo comparator
  Arms: normal saline

SUMMARY:
Purpose to evaluate the effects of topical tranexamic acid (TA) on reducing post-partum hemorrhage in pregnant women with hemorrhagic cesarean section

DETAILED DESCRIPTION:
Uterine atony is the major cause of postpartum hemorrhage (PPH), accounting for up to 80% of PPH cases. PPH is the leading cause of maternal morbidity and mortality worldwide, resulting in up to 28% of maternal deaths. Therefore, inducing a rapid and effective uterine contraction following delivery is an important issue. The aim of the study is to To explore the efficacy and safety of temporary uterine packing combined with topical tranexamic acid (TA) as an adjunct for reducing blood loss during a hemorrhagic cesarean delivery (CD), compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* patients who were admitted for an elective or non-emergency CS during labor and exposed to intraoperative bleeding about 800 ml

Exclusion Criteria:

* placenta praevia and placental abruption
* Women with a medical disorder,
* placenta accrete,
* allergy to TA, and
* intraoperative bleeding thanks to causes aside from uterine atony
* Patients over 40 or who have

  * pre-existing coagulation disorders,
* with a severe medical disorder
* allergy to tranexamic acid
* refuse to consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — patients who were admitted for an elective or non-emergency CS during labor and exposed to intraoperative bleeding about 800 ml
Enrollment: 180 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
number of patients need of additional pharmacological uterotonic | 24 hours post operative
  calculation number of patients need of additional pharmacological uterotonic

SECONDARY OUTCOMES:
estimation of intraoperative blood loss (ml) | during the operation
  measure Intraoperative blood loss in ml by gravimetric methods
amount of postoperative blood loss | 4 hours postoperative
  measure amount of blood loss post operative in ml by gravimetric methods
number of patient with postpartum hemorrhage | 24 hours post operative
  calculation of the number of the patients with blood loss >1000 ml

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided